CLINICAL TRIAL: NCT06489483
Title: Revealing the Action Regulation Mechanisms in the Human Brain
Brief Title: Action Regulation Behavioral
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of California, Riverside (Other)
Responsible Party: Principal Investigator, Nader Pouratian, Professor and Chair of Neurological Surgery, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU-2022-0555
Record Dates: First submitted 2024-06-26; First posted 2024-07-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Levodopa medication; motor cortex; basal ganglia
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's Disease Patients (Experimental): Patients that have been diagnosed with Parkinson's Disease and are responsive to levodopa medication. Patients will complete a behavioral task.
  Interventions: Behavioral: Action Regulation Movement Task
- Healthy Controls (Active Comparator): Men and women between the ages of 18-80. Spouse of PD patient who participates in this study with no history of any diagnosed neurological disease(s), including movement disorders or cognitive decline. No vision or hearing problems that impair ability to participate with the proposed tasks as assessed by the study investigators.
  Interventions: Behavioral: Action Regulation Movement Task

INTERVENTIONS:
Behavioral: Action Regulation Movement Task — A joystick is utilized to trace the movement of a visual stimulus on a computer screen. In stop signal task, the subjects are required to move a reference dot to reach to a target dot by controlling a joystick and stop their movements when the target turns red. During the switch task, subjects will be required to switch their joystick movement trajectory when the target location is switched to one of the other target locations.

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disorder involving a part of the brain that is responsible for motor control, which not only results in changes or disruptions in movement, but also cognitive dysfunctions. Given that the decline of muscle control such as tremors, with difficulty walking or the ability to switch tasks once in movement, greatly affects the quality of daily life. Action regulation is a critical executive function (cognitive control over behavior), which includes actions such as suppressing activity when selecting between options, making decisions about stopping unwanted or inappropriate actions, and switching to new actions in response to environmental changes. Parkinson's disease (PD) has been shown to disrupt action inhibition which can be considered a measure to the progression of PD.

The purpose of this research study is to better understand the mechanism of action regulations in PD patients and how action regulations in PD can be improved using dopaminergic treatment, which is a drug that either releases or involves dopamine, which is a neurotransmitter involved in sending signals to nerve cells.

You are asked to participate in this research study because you are receiving a dopaminergic medication for treatment of your Parkinson's disease. There is currently no theory that integrates the mechanisms of action regulation into a unified framework, which this study aims to address. The researchers hope to learn more about the mechanisms of action regulation in PD patients and to help decrease action regulation disruptions in PD patients. This study will help characterize the motor behavior of PD patients.

ELIGIBILITY:
For Parkinson's Disease Patients:

Inclusion Criteria:

* Diagnosis of Parkinson's Disease by a movement disorder neurologist
* Levodopa responsive with clearly defined "on" periods, with at least 30% improvement in UPDRS III scores on vs off
* Willingness and ability to complete the behavioral experiments for up 3.5 hours
* No vision or hearing problems that impair ability to participate with the proposed tasks as assessed by the study investigators

Exclusion Criteria:

* Patients with history of secondary Parkinsonism, stroke, or progressive central nervous system disease other than Parkinson's Disease
* Patients with a disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocol including cognitive decline, diagnosed forms of dementia, significant memory impairment (MoCA<23), or hearing loss that prevents adequate communication with researcher

For Healthy subjects:

Inclusion Criteria:

* No history any diagnosed neurological disease(s), including movement disorders or cognitive decline
* No vision or hearing problems that impair ability to participate with the proposed tasks as assessed by the study investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Stop-Signal Task | Baseline
  Each patient will complete a joystick-based stop-signal task which assesses reaction time, stop reaction time, accuracy, and joystick traces.
Switch Task | Baseline
  Each patient will complete a joystick-based switch task which assess reaction time, switch reaction time, accuracy, and joystick traces.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Following data acquisition, de-identified data will be shared with research team at University of California, Riverside.